CLINICAL TRIAL: NCT03104803
Title: Long-term Paired Associative Stimulation as a Treatment for Incomplete Spinal Cord Injury of Non-traumatic Origin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Validia Rehabilitation Center (Unknown); University of Helsinki (Other)
Responsible Party: Principal Investigator, Anastasia Shulga, MD, PhD, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULD 8100014-2
Record Dates: First submitted 2017-04-01; First posted 2017-04-07 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Spinal Cord Diseases; Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Diseases; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long-term PAS (Experimental): The intervention is given to one hand only
  Interventions: Device: long-term paired associative stimulation
- No intervention (No Intervention): Contralateral hand of the same patient

INTERVENTIONS:
Device: long-term paired associative stimulation — Paired associative stimulation (PAS) administered several times per week for 6 weeks to one hand. PAS comprises transcranial magnetic stimulation (eXimia magnetic stimulator, Nexstim Ltd, Helsinki, Finland) and peripheral nerve stimulation (given with Dantec Keypoint® electroneuromyography device (Natus Medical Incorporated, Pleasanton, CA, USA)).
  Arms: Long-term PAS

SUMMARY:
The investigators have recently shown in incomplete SCI patients that long-term paired associative stimulation is capable of restoring voluntary control over some paralyzed muscles and enhancing motor output in the weak muscles (1). In this study, the investigators will administer long-term paired associative stimulation to patients with incomplete SCI of non-traumatic origin.

ELIGIBILITY:
Inclusion Criteria:

* incomplete SCI of non-traumatic origin

Exclusion Criteria:

* epilepsy
* metal inclusion in the head area
* pacemaker
* hearing device
* high intracranial pressure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-05-27 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Daniels and Worthingham's Muscle Testing | 2 days after the last stimulation session
  each hand muscle is evaluated on 0-5 scale
Daniels and Worthingham's Muscle Testing | 1 month after the last stimulation session
  each hand muscle is evaluated on 0-5 scale

CONTACTS AND LOCATIONS:
Locations (1):
- BioMag laboratory, Helsinki, Finland

REFERENCES:
- [Result] Tolmacheva A, Savolainen S, Kirveskari E, Brandstack N, Makela JP, Shulga A. Paired associative stimulation improves hand function after non-traumatic spinal cord injury: A case series. Clin Neurophysiol Pract. 2019 Aug 13;4:178-183. doi: 10.1016/j.cnp.2019.07.002. eCollection 2019. PMID 31886442